CLINICAL TRIAL: NCT00051987
Title: A Randomized, Multicenter, Open-Label, Phase 2b Study of VELCADE Alone and VELCADE Plus Irinotecan in Patients With Relapsed or Refractory Colorectal Carcinoma
Brief Title: Phase 2b Study of VELCADE Alone and VELCADE Plus Irinotecan in Patients With Relapsed or Refractory Colorectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M34102-049
Record Dates: First submitted 2003-01-21; First posted 2003-01-22 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bortezomib; WW Domain-Containing Oxidoreductase

INTERVENTIONS:
Drug: VELCADE TM (bortezomib) for Injection, or PS-341

SUMMARY:
The purpose of this study is to evaluate how tumors in patients with colorectal carcinoma respond to treatment with VELCADE alone versus VELCADE given with irinotecan, and also to see what effects (good and bad) it has on you and your cancer.

DETAILED DESCRIPTION:
In this study, patients with colorectal cancer that is no longer responding to standard medical treatment with irinotecan or an irinotecan containing treatment will be randomized to treatment with VELCADE alone or to treatment with VELCADE in combination with irinotecan.

ELIGIBILITY:
Inclusion Criteria

* Patient has histologically confirmed inoperable locally advanced or metastatic CRC.
* Patient has measurable disease.
* Patient is not considered a candidate for immediate curative resection.
* Patient has received no more than 2 prior treatment regimens for metastatic disease, one of which must have contained irinotecan.
* Patient has relapsed or progressed while receiving an irinotecan-containing regimen.
* Patient has KPS of 70% or greater.
* Patient has a life expectancy greater than 3 months.
* Patient is 18 years of age or older.
* Female patient is postmenopausal, surgically sterilized, or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male patient agrees to use an acceptable method of birth control for the duration of the study.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to his or her future medical care.
* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.

Exclusion Criteria

* Patient has greater than or equal to Grade 2 neuropathy as defined by the NCI Common Toxicity Criteria (CTC):

  * Grade 2: Objective sensory loss or paresthesia (including tingling), interfering with function, but not interfering with activities of daily living (ADL).
  * Grade 3: Sensory loss or paresthesia interfering with ADL.
  * Grade 4: Permanent sensory loss that interferes with function.
* Patient has previously received treatment with VELCADE.
* Patient has other malignancies except non-melanoma skin cancers and carcinoma of the cervix in situ.
* Patient has received chemotherapy within 4 weeks prior to enrollment.
* Patient has received radiation therapy within 4 weeks prior to enrollment.
* Patient has received monoclonal antibodies within 6 weeks prior to enrollment.
* Patient had major surgery within 4 weeks prior to enrollment.
* Patient has inadequate organ function at Baseline (ie, Day 1 of Cycle 1) as defined by the following laboratory values:

  * Platelet count ≤ 100,000 x 109/L
  * Hemoglobin ≤ 8.0 g/dL
  * Absolute neutrophil count (ANC) ≤ 1.5 x 109/L
  * Aspartate transaminase (AST) ≥ 3 times the upper limit of the normal range (ULN)
  * Alanine transaminase (ALT) ≥ 3 times ULN
  * Total bilirubin ≥ 1.5 times ULN, unless clearly related to the disease
  * Calculated or measured creatinine clearance ≤ 60 mL/minute.
* Patient has had a myocardial infarction within 6 months of enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiogram (ECG) abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has symptomatic brain metastases.
* Patient has an active systemic infection requiring treatment.
* Patient has a history of inflammatory bowel disease.
* Patient has a history of allergic reaction attributable to compounds containing boron or mannitol.
* Patient previously required premature discontinuation of irinotecan therapy because of drug-related toxicity.
* Patient is known to be human immunodeficiency virus (HIV)-positive. Patients assessed by the investigator to be at risk for HIV infection should be tested in accordance with local regulations.
* Patient is known to be hepatitis B surface antigen-positive or has known active hepatitis C infection. Patients assessed by the investigator to be at risk for hepatitis B or C infection should be tested in accordance with local regulations.
* Patient has poorly controlled hypertension, diabetes mellitus, or another serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Female patient is pregnant or breast-feeding. Confirmation that the patient is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during the Screening period. Pregnancy testing is not required for postmenopausal or surgically sterilized women.
* Patient currently is enrolled in another clinical research study or has received an investigational agent for any reason within 4 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175
Dates: Start 2002-12; Primary Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Cooper Green Hospital / Jefferson Clinic P.C., Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Arkansas Cancer Center, Pine Bluff, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkley, California
  - California Cancer Center, Greenbrae, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - City of Hope Medical Group, Pasadena, California
  - H. Lee Moffit Cancer Center, Tampa, Florida
  - Rush Cancer Institute, Chicago, Illinois
  - Kentuckiana Cancer Institute, PLLC, Louisville, Kentucky
  - West Michigan Regional Cancer and Blood Center, Ludington, Michigan
  - Bond Clinic Inc., Rolla, Missouri
  - Nevada Cancer Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University, New York, New York
  - St. Lukes Rossevelt Hospital, New York, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health Sciences, Portland, Oregon
  - Memphis Cancer Center, PC, Memphis, Tennessee
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas